CLINICAL TRIAL: NCT03912090
Title: Using, Efficacity and Safety of Intranasal Fentanyl for the Treatment of Acute Severe Pain on the Pediatric Emergency Department of Mercy Hospital.
Brief Title: Intranasal Fentanyl for the Treatment of Acute Severe Pain on the Pediatric Emergency Department of Mercy Hospital.
Acronym: FENTANYLIN
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Régional Metz-Thionville (Other)
Responsible Party: Sponsor
Other Study IDs: 2018-07Obs-CHRMT
Record Dates: First submitted 2019-04-10; First posted 2019-04-11 (Actual); Last update posted 2019-05-14 (Actual); Status verified 2019-04

CONDITIONS: Acute Pain
Keywords: pediatric; fentanyl; intranasal; emergency
MeSH Terms: conditions — Acute Pain; Emergencies

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The treatment of acute severe pain in pediatric emergencies required a quick and effective therapeutic support. Actually in France, only peripheral venous access or oral therapies with onset of action are commonly used and only few treatments can be used to manage the acute severe pain in children. In June 2017, an intranasal fentanyl use protocol has been established in the pediatric emergency department of Mercy hospital-Metz. The intranasal fentanyl treatment has proved his effectiveness and safe condition in many countries since few years even though has not yet obtained a marketing authorization for use in children in France. In view of the information, parental permission was obtained before the intranasal administration. The efficacy and surveillance data in all patient records of children who benefited this analgesic protocol were retrospectively collected between June 2017 and August 2018. This retrospective study wants to describe the efficacy and safety of intranasal fentanyl on the pediatric emergency department.

ELIGIBILITY:
Inclusion Criteria:

* All patients who received fentanyl intranasal between june 2017 and august 2018

Exclusion Criteria:

* Lack of surveillance data in the medical record of the patient

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: * Pediatric patients of the emergency pediatric department of Mercy hospital
  * Coming for acute severe pain : EVA or FLACC scale >=6 for less than 6 hours
  * Age more than 12months
  * Weight 10kg to 68kg
  * Veinous access difficult to obtain
  * No contra-indication for fentanyl use
  * No contra-indication for intranasal administration
Sampling Method: Non-Probability Sample
Enrollment: 83 (Actual)
Dates: Start 2018-10-30 (Actual); Primary Completion 2019-04-01 (Actual); Study Completion 2019-05-01 (Actual)

PRIMARY OUTCOMES:
Pain scale evolution | Day 1
  Face Legs Activity Cry Consolability (FLACC) scale or Visual Analog Scale (VAS) FLACC scale involve, as its name implies, 5 items: face, legs, activity, cry and consolability with a score ranging from 0 to 2 each, knowing that 0 represents "no pain". The sum of each items is from 0 to 10, and 10 constitutes an intense pain.
  VAS is a 100-mm long horizontal line with verbal descriptors at each end to express the extremes of the feeling. Patients should mark the point on the line that the best correspond to their symptom severity. The patient's mark indicates pain severity and it's quantified by measuring the distance in millimeter from 0 (0 representes "no pain" and 100 represents "worst possible pain")

SECONDARY OUTCOMES:
Respiratory frequency | Day 1
  Respiratory frequency
Cardiac frequency | Day 1
  Cardiac frequency
Glasgow Coma scale | Day 1
  The Glasgow Coma scale (GCS) describes the level of consciousness. The GCS measures 3 functions: eye opening (with score between 1 and 4), verbal response (with score between 1 and 5) and motor response (with score between 1 and 6). Then, the sum of the scores is calculated. Pediatric brain injury are classified by severity 8 or lower reflecting the most severe, 9-12 being a moderate injury and 13-15 indicating a mild traumatic brain injury.
Oxygen saturation | Day 1
  SpO2

CONTACTS AND LOCATIONS:
Locations (1):
- CHR Metz Thionville, Metz, Moselle, France

IPD SHARING:
Plan to Share IPD: No